CLINICAL TRIAL: NCT07395193
Title: A Prospective Observational Study Comparing BiZact™, Coblation, and Bipolar Tonsillectomy Techniques
Brief Title: Comparative Evaluation of BiZact™, Coblation, and Bipolar Tonsillectomy Techniques
Acronym: BCB-Tonsillect
Status: Completed | Type: Observational
Sponsor: Medicana Bursa Hospital (Other)
Responsible Party: Principal Investigator, Oktay Bulut, Principal Investigator, Medicana Bursa Hospital
Other Study IDs: 2024/2
Record Dates: First submitted 2026-01-27; First posted 2026-02-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Tonsil Disease; Tonsil Disorder
Keywords: tonsillectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BiZact Tonsillectomy: Patients undergoing tonsillectomy using the BiZact™ device.
- Coblation Tonsillectomy: Patients undergoing tonsillectomy using the coblation technique.
- Bipolar Tonsillectomy: Patients undergoing tonsillectomy using bipolar electrocautery.

SUMMARY:
This prospective, non-randomized observational study compared the surgical outcomes of BiZact™, Coblation, and Bipolar tonsillectomy techniques in pediatric and adult patients. Operative efficiency, postoperative pain, recovery parameters, postoperative bleeding, and device-related costs were evaluated.

DETAILED DESCRIPTION:
Tonsillectomy is a commonly performed surgical procedure in otorhinolaryngology, and various techniques have been developed to improve operative efficiency and postoperative recovery. This prospective, non-randomized observational study included 150 patients aged 5-40 years who underwent tonsillectomy between November 2024 and September 2025. Patients were allocated to Bipolar, Coblation, or BiZact tonsillectomy groups based on surgeon preference and device availability.

Primary outcome measures were operative time and postoperative pain assessed using the visual analogue scale on postoperative days 1, 3, and 7. Secondary outcomes included time to first solid food intake, length of hospital stay, postoperative bleeding, bleeding management, and device-related cost. The study aimed to compare clinical outcomes, recovery profiles, and procedural efficiency among the three tonsillectomy techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 40 years
* Undergoing tonsillectomy
* Indication for surgery due to recurrent tonsillitis or obstructive sleep-related symptoms

Exclusion Criteria:

* Known coagulation disorders
* Presence of peritonsillar abscess
* Presence of craniofacial syndromes
* Incomplete follow-up data

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric and adult patients undergoing tonsillectomy at a tertiary care center.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Postoperative pain (Visual Analog Scale score) | Postoperative days 1, 3, and 7
  Postoperative pain was assessed using the Visual Analog Scale (VAS), a 10-cm scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Higher scores represent greater pain intensity.
Surgery time | During surgery

SECONDARY OUTCOMES:
Time to first solid food intake | Within the first postoperative week
Length of hospital stay | Postoperative Day 1
  Duration of hospitalization measured in days following tonsillectomy.
Postoperative bleeding | Up to 30 days postoperatively
Device cost per case | Perioperative period (day of surgery)
  Cost of the surgical device used for tonsillectomy, calculated per patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Medicana Bursa Hospital, Nilufer, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bulut O, et al. Comparative Evaluation of BiZact™, Coblation, and Bipolar Tonsillectomy Techniques. Unpublished data.